CLINICAL TRIAL: NCT06166914
Title: Evaluation of 5-fluorouracil and Low Molecular Weight Heparin Intraoperative Infusion in Preventing Proliferative Vitreoretinopathy in High Risk Pediatric Rhegmatogenous Retinal Detachment
Brief Title: Efficacy of 5-fluorouracil and Low Molecular Weight Heparin in High-risk Pediatric Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9163209
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Retinal Detachment; Proliferative Vitreoretinopathy
Keywords: pediatric retinal detachment; proliferative vitreoretinopathy; 5-Fluorouracil; Low molecular weight heparin
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial of patients enrolled sequentially into group A (treatment) and group B (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Group A received intraoperative infusion of 5-FU (200 µg/ml) and LMWH (5 IU/ml) during pars plana vitrectomy and silicone oil injection with scleral buckle in children under 14 years of age with high-risk PRRD
  Interventions: Drug: Intraoperative infusion of 5-FU (200 µg/ml) and LMWH (5 IU/ml)
- Control group (Placebo Comparator): Group B received infusion of normal saline during pars plana vitrectomy and silicone oil injection with scleral buckle in children under 14 years of age with high-risk PRRD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intraoperative infusion of 5-FU (200 µg/ml) and LMWH (5 IU/ml) — After informed consent, children under 14 years of age with high-risk PRRD underwent pars plana vitrectomy and silicone oil injection with scleral buckle divided into 2 groups in prospective randomized trial. Group A received intraoperative infusion of 5-FU (200 µg/ml) and LMWH (5 IU/ml).
  Arms: Treatment group
Drug: Placebo — After informed consent, children under 14 years of age with high-risk PRRD underwent pars plana vitrectomy and silicone oil injection with scleral buckle divided into 2 groups in prospective randomized trial. Group B received infusion of normal saline.
  Arms: Control group

SUMMARY:
EVALUATION OF 5-FLOUROURACIL AND LOW MOLECULAR WEIGHT HEPARIN INTRAOPERATIVE INFUSION IN PREVENTING PROLIFERATIVE VITREORETINOPATHY IN HIGH RISK PEDIATRIC RHEGMATOGENOUS RETINAL DETACHMENT

DETAILED DESCRIPTION:
After informed consent, children under 14 years of age with high-risk PRRD underwent pars plana vitrectomy and silicone oil injection with scleral buckle divided into 2 groups in prospective randomized trial. Group A received intraoperative infusion of 5-FU (200 µg/ml) and LMWH (5 IU/ml), group B received infusion of normal saline. Primary outcome was occurrence of recurrent PRRD within 12 weeks, secondary outcomes were occurrence of PVR, best corrected visual acuity (BCVA), number and timing of secondary procedures within 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Children under 14 years of age with RRD undergoing primary repair Preoperative PVR grade B or higher High risk RRD: uveitis; large, giant, or multiple tears; vitreous hemorrhage; preoperative choroidal detachments; aphakia; and large detachments involving greater than two quadrants of the eye

Exclusion Criteria:

Children with RRD related to penetrating ocular trauma involving the posterior segment Previous RD repair surgery Uncontrolled glaucoma or other concomitant ocular morbidities Patients with bleeding diathesis, hepatic and renal failure Corneal opacity sufficient to impair surgical view No light perception vision Inability to complete follow-up

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Recurrent RD due to PVR | 12 weeks post operative
  Clinical retinal detachment with any grade PVR

SECONDARY OUTCOMES:
Post operative PVR | 12 weeks post operative
  Any grade or degree of PVR at 6 and 12 weeks in accordance with the updated classification of PVR of the Retina Society (1991).
Best corrected visual acuity | 12 weeks post operative
  BCVA measured by Landolt's broken ring or illiterate E charts within 6 and 12 weeks in cooperative children.
Secondary procedures | 12 weeks post operative
  Number and extent of surgical procedures necessary to achieve retinal re-attachment within 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nasr M, Abdelhadi A, Bessa A, Ibrahim TM. Efficacy of 5-fluorouracil (5-FU) and low molecular weight heparin (LMWH) in high-risk pediatric retinal detachment; randomized clinical trial. BMC Ophthalmol. 2024 Mar 4;24(1):97. doi: 10.1186/s12886-024-03362-4. PMID 38433191